CLINICAL TRIAL: NCT06393894
Title: A Prospective Registry to Assess Atherosclerosis Risk Factors and Their Relationship With Coronary Plaque Properties and Genetic Variations in Patients With Early Atherosclerosis of Unclear Origin.
Brief Title: Latvian Early Atherosclerosis Registry
Status: Recruiting | Type: Observational
Sponsor: Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Principal Investigator, Karlis Trusinskis, Professor, Pauls Stradins Clinical University Hospital
Other Study IDs: AAR-0419
Record Dates: First submitted 2020-09-15; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Atherosclerosis, Coronary
Keywords: Coronary artery disease; Early atherosclerosis; MicroRNA; Near infrared spectroscopy
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Spectroscopy, Near-Infrared; Genetic Testing; Apolipoproteins B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Near infrared spectroscopy — Near infrared spectroscopy (NIRS) is an intravascular imaging technique. Patients after coronary angiography with or without angioplasty will undergo NIRS if deemed suitable by the interventionalist. NIRS has a high sensitivity and specificity for lipid core plaque detection.
Genetic: Genetic testing for LDLR, APOB, PCSK9 and LDLRAP1 mutations and niR-126, -145 and -155 expression. — Patients without explicit atherosclerosis risk factors and known genetic disorders will undergo genetic testing for LDLR, APOB, PCSK9 and LDLRAP1 genes in order to evaluate the presence of gene variations as a cause for early atherosclerosis. MiRNA-126, -145 and -155 expression in patients serum samples will be evaluated and correlated with plaque lipid core in near infrared spectroscopy (NIRS) imaging.

SUMMARY:
Atherosclerosis and its complications are a global problem. There are several widely known and proven risk factors that promotes atherogenesis in the majority of patients. However, significant proportion of apparently healthy and young patients with cardiovascular disease but yet without recognized atherogenesis promoting risk factors can be observed in clinical practice. It highlights the need of new risk markers for early atherosclerosis diagnostics to prevent serious cardiovascular complications in these patients and in population in general. The interest in the negative impact of genetic variance, gene regulation on atherogenesis is growing. Therefore the purpose of this study is to analyze the impact of genetic variance and microRNA expression on early atherosclerosis development in the population of young, apparently healthy patients with coronary atherosclerosis. The primary hypothesis is that the group of patients with premature atherosclerosis have common genetic variations promoting early atherosclerosis development. The secondary hypothesis is that specific circulating microRNA expression (miR-126, miR-145 and miR-155) correlate with plaque lipid core by near infrared spectroscopy (NIRS) analysis.

DETAILED DESCRIPTION:
Patients with early atherosclerosis undergoing coronary angiography or percutaneous transluminal coronary angioplasty (PTCA) at Pauls Stradins Clinical University Hospital, Latvia will be included in the early atherosclerosis registry. Patients without explicit atherosclerosis risk factors undergoing coronary angiography or PTCA will undergo near-infrared spectroscopy imaging and blood samples for microRNA expression evaluation and genetic analysis will be obtained.

Exclusion criteria:

* Refusion to participate in the registry
* Men ≥55 years and women ≥65 years
* Coronary artery atherosclerosis < 50% or ≥50% without proven ischaemia and planned revascularization or no history of coronary artery revascularization

Exclusion criteria for additional genetic analysis and intravascular coronary imaging:

* Diabetes mellitus
* Serum total cholesterol ≥ 7 mmol/l and/or LDL ≥ 5 mmol/l
* Family hypercholesterolemia
* Positive family history of cardiovascular disease (myocardial infarction, sudden cardiac death or cardiovascular disease of first-degree relatives at a young age - men <55 years, women <65 years)
* ≥20 pack years of smoking
* Malignant or resistant hypertension ≥ 10 years
* Body mass index ≥40 kg/m2

At the time of recruitment demographic characteristics, medical and family history, anthropometric parameters, smoking status, history of other risk factors and daily used medications will be recorded and venous blood samples will be obtained.

In obtained venous blood samples study researchers will evaluate biochemistry analysis which includes high-density and low-density lipoprotein cholesterols, total cholesterol, triglycerides, alanine aminotransaminase, aspartate aminotransferase, bilirubin, creatine kinase, glucose and glycated haemoglobin levels. Genetic analysis will include sequencing of the four major candidate genes for monogenic hypercholesterolemia (LDLR, APOB, PCSK9 and LDLRAP1). microRNA (miR)-126, miR-145 and miR-155 expression will be evaluated in all venous blood samples.

Patients undergoing repeated coronary angiography or PTCA will undergo intravascular imaging - near-infrared spectroscopy to determine coronary plaque lipidic tissue content.

Follow-up phone calls will be performed after 6, 12 and 24 months. In the follow-up study researchers will obtain additional information on study participants including smoking status, daily used medications and anthropometric parameters.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent
* Early atherosclerosis defined as coronary atherosclerosis in men aged <55 years and women <65 years
* Coronary artery atherosclerosis with angiographically proven coronary vessel luminal stenosis ≥ 50% and ischaemia
* Coronary artery atherosclerosis with planned revascularization
* History of coronary artery revascularization (PTCA or coronary artery bypass surgery)
* Coronary vessel suitable for NIRS pullback

Exclusion criteria:

* Diabetes
* Total cholesterol ≥7 mmol/l and/or LDL ≥ 5 mmol/l
* family hypercholesterolemia
* positive family history of early cardiovascular disease (myocardial infarction, sudden cardiac death or cardiovascular disease of first degree relatives at young age - men <55 years, women <65 years)
* malignant or resistant hypertension ≥ 10 years
* body mass index ≥40 kg/m 2 )
* 20 or more pack years of smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to coronary angiography with or without angioplasty meeting the inclusion criteria and without explicit exclusion criteria will be screened for this registry.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Genetics | 12 months
  Correlation between intravascular plaque characteristic data and gene variations in LDLR (low density lipoprotein receptor), APOB (Apolipoprotein B), PCSK9 (proprotein convertase subtilisin/kexin type 9) and LDLRAP1 (Low Density Lipoprotein Receptor Adaptor Protein 1).

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 12 months
  Composite of nonfatal myocardial infarction, cardiovascular death, repeat coronary revascularization
Intravascular coronary imaging | 12 months
  Intravascular plaque characteristic assesment by intravascular diagnostic modalities (intravascular ultrasound and/or near infrared spectroscopy).
Target lesion revascularization | 12 months
  Revascularization post-stenting within the stent or within the 5-mm borders adjacent to the stent

CONTACTS AND LOCATIONS:
Locations (1):
- Pauls Stradins Clinical University hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No